CLINICAL TRIAL: NCT06841601
Title: Effectiveness of Vibratory Versus Cold Stimuli on Pain Perception During Needle Insertion in Children
Brief Title: Effectiveness of Vibratory Versus Cold Stimuli on Pain Perception in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Dina Sharaf, Lecturer of Pediatric Dentistry, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0568-12/22
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Pain Perception
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- topical anesthesia (Active Comparator): Topical anesthetic gels are applied prior to injection at the injection site to minimize pain upon insertion of the needle during local anesthesia
  Interventions: Other: topical anesthetic gel
- vibration (Experimental): Vibration using a vibrating devise (Buzzy) can help reduce the pain during local anesthesia injection. It is placed extra-orally before and during needle insertion
  Interventions: Other: Vibration
- cold pack (Experimental): Cold pack provided with the Buzzy device will be used without the vibration mode of the device. It is applied extra-orally before and during needle insertion.
  Interventions: Other: Cold pack

INTERVENTIONS:
Other: topical anesthetic gel — gels applied directly to the mucous membranes to provide localized relief of pain by numbing the area. They typically contain active ingredients such as lidocaine, benzocaine, or prilocaine, which work by blocking nerve signals to reduce sensation and discomfort
  Arms: topical anesthesia
Other: Vibration — The vibration generated by the Buzzy device functions as a non-pharmacological agent that can reduce pain perception in children based on the principles of the Gate Control Theory of Pain.
  Arms: vibration
Other: Cold pack — cold packs are also provided by the Buzzy device. they act as non-pharmacological agents that can reduce pain perception in children based on the Gate Control Theory of Pain.
  Arms: cold pack

SUMMARY:
Local anesthesia is an anxiety-provoking procedure. Pain control is important for effective behavior guidance, specially among pediatric patients.

This study aims to evaluate the effectiveness of Buzzy® as a topical anesthetic in pain perception through two ways: once using vibration mode without the cold pack and the other using the cold pack without vibration and comparing it to topical anesthetic gel during different anesthetic techniques Methods: A randomized controlled clinical trial involving 72 healthy cooperative patients aged 5-9 years. They will be allocated to receive local anesthesia either using the vibration mode of Buzzy Bee (test group) or the cold pack of Buzzy Bee (test group) or conventional topical anesthetic gel (control group). Pain response will be assessed using Visual Analog Scale (VAS) and SEM scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated for simple restorative procedures.
2. Children with physical status ASA I, II.
3. Children with no learning disabilities
4. Positive or definitely positive behavior during preoperative assessments according to the Frankl Scale.
5. Patients whom parents will give consent to participate

Exclusion Criteria:

1. Patients allergic to local anesthesia or having a family history of allergy to local anesthesia.
2. Patients with acute oral or facial infection (swelling and/or cellulites)
3. Having active sites of pathosis in the area of injection that could affect anesthetic assessment.
4. Children with special health care needs.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-02-23 (Estimated); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Pain perception during needle insertion in different anesthetic techniques Using SEM scale | during the procedure (needle insertion)
  Objective method of pain assessment using SEM (sound, eye and movement scale). It is a behavioral assessment tool to evaluate pain and distress responses in children during dental procedures. It uses scores from 0 till 3 according to increasing levels of distress.

SECONDARY OUTCOMES:
Pain will be assessed after local anesthesia injection by means of Visual analogue scale. | immediately after the procedure (needle insertion)
  Subjective method of pain assessment where patients will be instructed how to point to the position on the line between faces to indicate how much pain they felt during local anesthesia administration. The total scores range from 0 to 10. Happy to sad faces are connected to the line, with a higher score indicating more severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided